CLINICAL TRIAL: NCT01878188
Title: Phase I Study of BC-819/PEI and BCG in Patients With Superficial Transitional Cell Bladder Carcinoma
Brief Title: Pilot Study of BC-819/PEI and BCG in Patients With Superficial Transitional Cell Bladder Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anchiano Therapeutics Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-BLAD-01
Record Dates: First submitted 2013-05-29; First posted 2013-06-14 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Transitional Cell Carcinoma of Bladder
Keywords: inodiftagene vixteplasmid
MeSH Terms: interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BC-819/PEI and BCG alternating (Experimental): 4 or 6 weekly treatments of BC-819/PEI alternating with 6 treatments of BCG
  Interventions: Drug: BC-819/PEI; Drug: BCG Vaccine
- BC-819/PEI and BCG Vaccine sequential (Experimental): 4 weekly treatments of BC-819/PEI followed by 6 weekly treatments of BCG
  Interventions: Drug: BC-819/PEI; Drug: BCG Vaccine
- twice-weekly treatments of BC-819 and BCG (Experimental): 6 twice-weekly treatments of BC-819/PEI and BCG
  Interventions: Drug: BC-819/PEI; Drug: BCG Vaccine

INTERVENTIONS:
Drug: BC-819/PEI — Intravesical instillation
Drug: BCG Vaccine — intravesical instillations
  Other Names: OncoTICE

SUMMARY:
* Safety and tolerability of three regimens of intravesically administered BC-819/PEI and BCG (number of participants with AEs, discontinuations due to AEs)
* Recurrence after treatment with BC-819/PEI and BCG
* Approximately 38 patients with superficial transitional cell carcinoma TCC) of the bladder
* After initial evaluation and qualification, patients will be randomized to one of three treatment groups, either alternating, sequential or twice weekly

ELIGIBILITY:
Inclusion Criteria:

1. Patients with superficial papillary transitional cell carcinoma of the bladder for whom BCG is clinically indicated. If CIS is present, diagnosis needs to be confirmed by biopsy prior to the start of the study.
2. Males or females more than 18 years old
3. All papillary tumors must be resected within 8 weeks prior to the start of study therapy.
4. ECOG performance status 2 or less.
5. Adequate hematologic function, as demonstrated by

   1. Hemoglobin 10 g/dL or higher
   2. ANC 1.5 x 109/L or higher
   3. Platelets higher than 100 x 109/L
6. Adequate liver and renal function as demonstrated by

   1. AST and ALT each 3.0 x ULN or less
   2. Total bilirubin 1.5 x ULN or less
   3. Creatinine 1.5 X ULN OR less, creatinine clearance >60 mL/min
7. If fertile and sexually active, must use adequate contraception
8. Must be able to comply with protocol requirements, including attendance at required clinic visits.
9. Patients must provide written informed consent.

   -

Exclusion Criteria:

1. Patients who are candidates for either partial or total bladder resection, unless either medically contraindicated or who have refused surgery.
2. Patients with a tumor in a diverticulum, in the prostatic urethra, or covering the ureteral orifice.
3. Patients who have received cytotoxic drugs, systemic corticosteroids or any investigational drug for any indication within 4 weeks of the start of protocol treatment.
4. Patients who have received any intravesical therapy other than surgical resection within 8 weeks prior to the start of protocol treatment.
5. Patients who have received radiation therapy for bladder cancer at any time or for any condition within 4 months prior to the start of protocol treatment.
6. Patients who have active infections, including urinary tract infections, whether viral, bacterial or fungal and requiring therapy.
7. Patients who are receiving coumadin.
8. Patients who have had to discontinue a past course of BCG due to toxicity.
9. Patients who are having urinary tract signs or symptoms from recent urinary tract procedures or manipulations, such as biopsies or catheterizations.
10. Patients who are known to be HIV positive.
11. Females who are pregnant or breast feeding.
12. Presence of any medical, psychological or social condition or situation which may, in the investigator's opinion, make it difficult for the patient to tolerate study medication or comply with study procedures and other requirements. This includes but is not limited to active infections, poorly controlled diabetes, uncontrolled cardiac arrhythmias, angina pectoris, or hypertension.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of three regimens of intravesically administered BC-819/PEI and BCG by number of subjects with AEs and change from baseline for clinical safety laboratory tests | 3 months

SECONDARY OUTCOMES:
Recurrence of bladder cancer after treatment with BC-819/PEI and BCG | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ami Sidi, MD, Principal Investigator — Wolfson Medical Center; Sarel Halachmi, MD, Principal Investigator — Bnai-Zion Medical Center, Haifa, Israel; Ilan Leibovitch, MD, Principal Investigator — Meir Medical Center, Kfar-Saba, Israel; Ofer Gofrit, MD, Principal Investigator — Hadassah Ein Karem Medical Center; Amnon Zisman, MD, Principal Investigator — Assaf Harofe Medical Center; Abraham Stein, MD, Principal Investigator — Carmel Hospital,Haifa; Haim Matzkin, MD, Principal Investigator — Tel Aviv Medical Center
Locations (7):
- Israel (7):
  - Bnai Zion MC, Haifa
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Ein Karem Medical Center, Jerusalem
  - Meir MC, Kfar Saba
  - Tel Aviv Medical Center, Tel Aviv
  - Assaf Harofe Medical Center, Ẕerifin

REFERENCES:
- See also: Related Info — http://www.biocancell.com/